CLINICAL TRIAL: NCT03974893
Title: Dietary Intake, Sarcopenic Obesity, and Other Treatment-Related Outcomes in Indian Children With Acute Lymphoblastic Leukemia: A Pilot Study
Brief Title: Dietary Intake, Sarcopenic Obesity, and Other Treatment-Related Outcomes in Indian Children With Acute Lymphoblastic Leukemia
Acronym: TATA
Status: Active, not recruiting | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Tata Memorial Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: AAAR8814
Record Dates: First submitted 2019-06-03; First posted 2019-06-05 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Sarcopenic Obesity
Keywords: Dietary intake; Diet; Acute lymphoblastic leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Diet, Vegetarian

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vegetarian Diet: Includes children following a vegetarian diet.
  Interventions: Other: Vegetarian Diet
- Non-Vegetarian Diet: Includes children following a non-vegetarian diet.

INTERVENTIONS:
Other: Vegetarian Diet — Dietary information will be collected utilizing a food record at four time points in therapy reflecting different intensities/drug exposures of treatment.
  Groups: Vegetarian Diet

SUMMARY:
Sarcopenic obesity occurs when there is a loss of muscle and gain of fat in the body. With this study, the investigators will explore how nutritional status at the beginning of the treatment can cause changes in your child's body fat compared to muscle in the body. The investigators will also look at how these changes can impact a child's cancer treatment, survival from treatment, and if there is any deterioration in health and nutrition status. The primary objective of this study is to establish the incidence of sarcopenic obesity, measured by dual-energy x-ray absorptiometry (DEXA), among Indian children and adolescents with acute lymphoblastic leukemia (ALL).

DETAILED DESCRIPTION:
Survival of childhood ALL exceeds 80% in an increasing number of many low-middle income countries (LMIC). Recent studies have found that the effects of obesity on survival are observed within the first several years of diagnosis, thus impacting immediate health outcome. Of concern is the developing body of evidence that the effects of obesity may be underestimated and its effect on outcome may be even more pronounced when it is defined by body composition. An elevated body mass index (BMI) can be comprised of increased fat-free mass (FFM) or fat-mass (FM) or a combination of both. Evidence suggests that an increase of FM is a stronger predictor of risk of chronic disease rather than BMI. The evaluation of FM and FFM appears to have clinical implications in both adult and pediatric oncology, particularly in patients with Sarcopenic Obesity (SO) (increased FM and reduced FFM). Among children with ALL located in both high income countries (HIC) and LMIC, remediation of poor nutritional status during treatment removes its adverse effect on survival at the end of treatment. targeting dietary patterns may be a more effective approach when considering dietary interventions. One plausible way to examine the association of dietary patterns with the development of SO in pediatric ALL is to compare a vegetarian diet to a non-vegetarian diet and investigate how they are associated with its development. Children and adolescents with ALL at Tata Memorial Center (TMC) are well suited for this investigation because at least 30% of children follow a vegetarian diet, are easily identified, and the diets are not interchangeable. The benefit of the proposed model eliminates the need for dietary intervention prior to the study, which will examine how SO, accumulation of FM and the loss of FFM, develops among children and adolescents with ALL adhering to a vegetarian compared to non-vegetarian diet. Additionally, this study will examine the interaction of physical activity and diet while considering influential variables on the development of SO.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with ALL
* Able to consume ≥ 80% of dietary requirements enterally
* Adequate performance status (Lansky score ≥70)
* Receiving standard treatment for ALL on or as per the Indian Childhood Collaborative Leukemia Group's protocol (ICiCLe).

Exclusion Criteria:

* Refusal of consent
* Relapsed ALL
* Down's syndrome; (Other congenital anomalies too)
* Therapy initiated elsewhere

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 100 eligible children aged 5 - 15 years old will be recruited at Tata Memorial Hospital in Mumbai, India. Any children with deteriorating health or not being able to perform diet and exercise routines are ineligible. Children getting therapy outside Tata are not eligible.
Sampling Method: Probability Sample
Enrollment: 115 (Actual)
Dates: Start 2019-04-18 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of Sarcopenic Obesity | 6 months
  Incidence of sarcopenic obesity, measured by dual-energy x-ray absorptiometry (DEXA), among Indian children and adolescents with ALL.

SECONDARY OUTCOMES:
Association of a Vegetarian Diet and Sarcopenic Obesity | 6 months
  Association of a vegetarian compared to a non-vegetarian diet and sarcopenic obesity, measured by dual-energy x-ray absorptiometry (DEXA)

CONTACTS AND LOCATIONS:
Overall Officials: Elena J. Ladas, PhD, RD, Principal Investigator — Columbia University
Locations (1):
- Tata Memorial Hospital, Mumbai, India

IPD SHARING:
Plan to Share IPD: No